CLINICAL TRIAL: NCT01991938
Title: A Phase I Dose Escalation Study of VS-5584, a Dual PI3K/mTOR Inhibitor, in Subjects With Advanced Non-Hematologic Malignancies or Lymphoma
Brief Title: Phase I Dose Escalation Study of VS-5584 in Subjects With Advanced Non-Hematologic Malignancies or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of recruitment and the company's decision to de-prioritize 5584 development
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-5584-101
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Non Hematologic Cancers; Metastatic Cancer; Lymphoma
Keywords: PI3K Inhibitor; mTOR Inhibitor; Dual PI3K/mTOR Inhibitor; CSC; Cancer Stem Cells
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma | interventions — VS-5584

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VS-5584 (Experimental): Oral VS-5584 administered once daily on Day 1, 3, 5, 8, 10, 12, 15, 17 and 19 of each cycle
  Interventions: Drug: VS-5584

INTERVENTIONS:
Drug: VS-5584

SUMMARY:
This is a Phase I, open-label, multicenter, dose-escalation trial of VS-5584, a PI3K/mTOR kinase inhibitor, in subjects with advanced non-hematologic malignancies or lymphoma. This clinical study is comprised of 2 sequential parts: Part 1 (Dose Escalation) and Part 2 (Expansion). The purpose of this study is to evaluate the safety (including the recommended Phase II dose), pharmacokinetics (the amount of VS-5584 in subject's blood) and the anti-cancer activity of VS-5584. Biomarkers (genes or proteins that may predict or show how subject's body may respond to VS-5584) will also be assessed in archival tumor tissue, tumor biopsies (in consenting subjects), and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed and dated informed consent prior to initiation of any study procedures.
2. Age ≥ 18 years.
3. Subjects must have a histopathologically confirmed diagnosis of an advanced non-hematologic malignancy or lymphoma or indolent NHL/CLL.
4. Subjects must have no alternate therapy of proven benefit or have refused standard therapy.
5. All clinically significant toxicities from prior chemotherapy must be ≤ Grade 1.
6. ECOG performance status of 0 or 1, measured at screening and immediately before the start of treatment.
7. Predicted life expectancy of ≥ 3 months.
8. Fasting blood glucose of ≤ 140 mg/dL (7.8 mmol/L).
9. Adequate renal function [creatinine ≤ 1.5x ULN (upper limit of normal)] or GFR of ≥ 60mL/min.
10. Adequate hepatic function (total bilirubin ≤ 1.5x ULN for the institution; AST [aspartate transaminase] and ALT [alanine transaminase] ≤ 3x ULN).
11. Adequate bone marrow function (hemoglobin ≥ 9.0 g/dL; platelets ≥ 75 x10^9 cells/L; absolute neutrophil count ≥ 1.0x10^9 cells/L).
12. Corrected QT interval (QTc) < 470 ms (as calculated by the Fridericia correction formula).
13. Negative pregnancy test for women of child-bearing potential.
14. Men and women of child bearing potential must agree to use adequate birth control throughout their participation in the study and for 60 days following the last study treatment.
15. Willing and able to participate in the trial and comply with all trial requirements.
16. Subjects must have archival tumor tissue available for mutational analysis. A study specific biopsy can be performed if archival tissue is not available.
17. Stable brain metastases either treated or being treated with a stable dose of steroids/ anticonvulsants, with no dose change within 28 days prior to the first dose of study drug, will be allowed.

Exclusion Criteria:

1. Gastrointestinal (GI) condition which could interfere with the swallowing or absorption of study medication.
2. Uncontrolled or severe concurrent medical condition including cardiovascular disease (e.g., myocardial infarct, unstable angina, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, cardiac amyloidosis, transient ischemic attacks, CVA, coronary artery or other vascular stents).
3. A past history of, or current uncontrolled hypertension. Blood pressure must be adequately controlled prior to dosing with VS-5584.
4. Prior history of a hypertensive reaction to a kinase inhibitor
5. History of upper gastrointestinal bleeding, ulceration, or perforation within 12 months prior to the first dose of study drug.
6. Subjects with known infection with human immunodeficiency virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS) (testing not required).
7. Subjects with known active Hepatitis A, B or C (testing not required).
8. Subjects being actively treated for a secondary malignancy.
9. Cancer-directed therapy (chemotherapy, radiotherapy, hormonal therapy with the exception of LHRH agonists for prostate cancer, biologic or immunotherapy, etc.) within 21 days of the first dose of study drug or 5 half-lives, whichever is shorter. Palliative radiotherapy is allowed prior to initiating treatment if associated toxicity resolved to ≤ Grade 1.
10. Subjects currently taking medications known to be strong CYP3A4 inhibitors.
11. Major surgery within 28 days prior to the first dose of study drug.
12. Subjects with acute or chronic pancreatitis.
13. Subjects with diabetes mellitus requiring insulin treatment or subjects with a HbA1C > 7.
14. Use of an investigational drug within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. A minimum of 14 days between termination of the investigational drug and administration of the study treatment is required. In addition, any drug-related toxicity except alopecia should have recovered to grade 1 or less.
15. Women who are pregnant or breastfeeding.
16. Any evidence of serious active infections.
17. Uncontrolled intercurrent illness involving any other organ system or a social situation that would, in investigator's opinion, place the subject at unacceptable risk, limit compliance, or confound interpretation of safety or other results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of VS-5584 in subjects with advanced non-hematologic malignancies or lymphoma | From start of treatment to end of treatment, an expected average of 6 weeks
  Serious Adverse events, Adverse events and their frequency, duration and severity, physical examination, laboratory parameters, vital signs and ECGs as determined based on CTCAE (Common Toxicity Criteria for Adverse Effects) V4.03. A Safety Monitoring Committee will review safety information.
Determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) and schedule of VS-5584 administered to subjects with advanced non-hematologic malignancies or lymphoma | From start of treatment to end of Cycle 1 (21 day cycles)
  The RP2D will be determined based on the MTD of VS-5584 as determined by number of participants with dose limiting toxicities related to VS-5584. Observations related to pharmacokinetics, pharmacodynamics, and any VS-5584 related toxicities may be included in the rationale supporting the RP2D and schedule and will not exceed the MTD.

SECONDARY OUTCOMES:
Assess the pharmacokinetics of VS-5584 | Time points on Day 1, 2, 3, 17, 18
  PK (pharmacokinetics) parameters, including but not limited to plasma concentration, clearance, AUC (Area Under Curve, 0-24 and 0-t), Cmax, Tmax, and T1/2

OTHER OUTCOMES:
Evaluate the efficacy of VS-5584 | Every 6 weeks to end of treatment, expected average of 6 weeks
  Response rate and progression-free survival as determined by Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1 or by the Revised Response Criteria for Malignant Lymphoma
Evaluate the time to new lesion | Expected average of 6 weeks from start of treatment to end of treatment
Evaluate duration of response to VS-5584 compared with duration of response to prior therapy | Expected average of 6 weeks from start of treatment to end of treatment
Examine the pharmacodynamic effect of VS-5584 on target proteins in platelet rich plasma and tumor biopsies | Platelet rich plasma time points: Day 1, 2, 8, 17; Tumor biopsies time points: Screening, Day 22, and at the time of progression
  Pharmacodynamic and predictive response biomarkers intended to demonstrate inhibition of the molecular target and determination of the mechanism of action will be assessed in archival tissue and tumor biopsies and platelet rich plasma samples.
Examine if tumor genetic alterations and/or plasma biomarkers correlate with response to VS-5584 therapy | start of treatment to end of treatment, an expected average of 6 weeks
  Tumor genetic alterations and/or plasma biomarkers compared with response to VS-5584, as determined by Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1 or Revised Response Criteria for Malignant Lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (5):
- United States (4):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
- The Royal Marsden, Sutton, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No